CLINICAL TRIAL: NCT06628024
Title: Determination of the Postprandial Amino Acid Uptake Kinetics of Yoghurt Vs Milk: a Randomized Controlled Clinical Trial in Health Individuals - a Bioavailability Study
Brief Title: Determination of the Postprandial Amino Acid Uptake Kinetics of Yoghurt Vs Milk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Nutraferm; 24REX0075382
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Amino Acids; Milk; Yoghurt
MeSH Terms: interventions — Milk; Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoghurt (Experimental): Yoghurt test product (Commercially available)
  Interventions: Other: Yoghurt
- Milk (Other): Commercially available product
  Interventions: Other: Milk

INTERVENTIONS:
Other: Milk — Milk
  Arms: Milk
Other: Yoghurt — Yoghurt
  Arms: Yoghurt

SUMMARY:
Subjects will visit the study site twice in a fasting state. Subjects asked to consume one of the two study products in a random order. Subjects will consume one serving of the study product (T = 0 minutes). Study product intake should take place within 10 minutes (+/-5 minutes). Blood samples will be taken at baseline and then at various timepoints after product intake. A follow up call will take place 7 days after the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 40 years at time of ICF signature
2. Body Mass Index (BMI) ≥ 18.5 and ≤ 27.0 kg/m2
3. Written informed consent
4. Willingness and ability to comply with the protocol
5. Judged by the Investigator to be in good health

Exclusion Criteria:

1. Any known ongoing medical condition that interferes significantly with absorption and digestion and/or gastrointestinal (GI) function (e.g. inflammatory bowel disease, gastroesophageal reflux disease, celiac disease, diaphragmatic hernia or diaphragmatic surgery, gastric ulcer, gastritis, gall bladder problems, pancreatitis, GI cancer, oesophageal and/or gastric surgery), in opinion of the investigator.
2. Known renal or hepatic diseases that may interfere with protein metabolism, including but not limited to acute hepatitis, chronic liver disease, nephritis, cystinuria, chronic kidney disease, in the opinion of the investigator.
3. Use of systemic medication within the past 3 weeks prior to screening which in the opinion of the investigator may influence gastric acid production and/or gastrointestinal motility or function and/or protein metabolism (for example: antibiotics, anticonvulsants, prokinetics, antacids, opioid analgesics, anticoagulants, corticosteroids, laxatives, growth hormone, testosterone, immunosuppressants, or insulin).
4. Known Diabetes Mellitus type I or type II, insulin resistance or metabolic syndrome.
5. Any ongoing cancer and/or cancer treatment (except for non metastasizing cancer e.g basal cell carcinoma).
6. Known anaemia or low haemoglobin or low iron status
7. Any known bleeding disorder.
8. Adherence to a strict dietary regime (e.g. vegetarian/ vegan/ paleo/ketogenic/ intermittent fasting/ high protein diet (>1.6 g/kg body weight/day) or a weight loss program.
9. Any known allergies or intolerances to ingredients of the study product, i.e. cow's milk allergies, lactose intolerance.
10. Known pregnancy and/or lactation.
11. Current smoking / vaping/ use of e-cigarette or stopped smoking for <

1 month prior to screening (except for incidental smoking of ≤ 3 cigarettes/ e-cigarettes/cigars/pipes per week on average in the last month prior to screening). 12. Average alcohol use of > 21 glasses per week for men or > 14 glasses per week for women (on average during the last 6 months prior to screening). 13. Drug or medicine abuse in opinion of the investigator. 14. Use of any nutritional supplements or additional protein supplements or nutritional support within 4 weeks prior to screening. 15. Known difficulties with placement of and/or blood drawings from a cannula. 16. Participation in any other clinical study with investigational or marketed products concomitantly or within four weeks before study visit

* Major medical or surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation relevant in the opinion of the investigator.
* Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.
* Employees of Danone Research and of the investigational site and/or their family members or relatives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Total amino acid concentrations after ingestion of product A vs B in 16 healthy adults | For 4 hours after product intake
  To compare the relative amount (iAUC) total amino acids (TAA) appearing in the blood for the 4-hour period after the ingestion of product A versus B.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) after ingestion of product A vs B in 16 healthy adults | For 4 hours after product intake
  To compare the maximum concentration (Cmax) and time to peak (Tmax) for total amino acids appearing in the blood for the 4-hour period after the ingestion of product A versus B in 16 healthy adults.

OTHER OUTCOMES:
Time to peak of essential amino acids after ingestion of product A vs B in 16 healthy adults | For 4 hours after product intake
  To compare time to peak (Tmax), for essential amino acids (EAA) of product A versus product B.
Relative amount of essential amino acid concentrations after consumption of product A vs. product B in 16 healthy adults. | For 4 hours after product intake
  To compare the relative amount (iAUC) of essential amino acids (EAAs) appearing in the blood for the 4-hour period after the ingestion of product A versus product B.
Maximum concentration (Cmax) of essential amino acids (EAAs) after product A vs. product B in 16 healthy adults. | For 4 hours after product intake
  To compare maximum concentration (Cmax) of essential amino acids (EAAs) appearing in the blood for the 4-hour period after the ingestion of product A versus product B.
Time to peak of leucine product A vs. product B in 16 healthy adults | For 4 hours after product intake
  To compare time to peak (Tmax) for leucine of product A versus product B.
Relative amount of leucine after product A vs. product B in 16 healthy adults. | For 4 hours after product intake
  To compare the relative amount (iAUC) of leucine appearing in the blood for the 4-hour period after the ingestion of product A versus product B.
Maximum concentration of leucine after product A vs. product B in 16 healthy adults | For 4 hours after product intake
  To compare maximum concentration (Cmax) of leucine appearing in the blood for the 4-hour period after the ingestion of product A versus product B.

CONTACTS AND LOCATIONS:
Locations (1):
- EB FlevoResearch, Almere Stad, Netherlands

IPD SHARING:
Plan to Share IPD: No